CLINICAL TRIAL: NCT07226271
Title: Consumer Perceptions of Alcoholic Beverages
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25-1870
Record Dates: First submitted 2025-11-03; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Natural Claim (Experimental)
  Interventions: Behavioral: Natural Claim
- Sugar Claim (Experimental)
  Interventions: Behavioral: Sugar Claim
- Fruit Claim (Experimental)
  Interventions: Behavioral: Fruit Claim
- No-claim Control (No Intervention)

INTERVENTIONS:
Behavioral: Natural Claim — Participants assigned to this condition will view three alcoholic beverages that carry the following claim: All natural flavors
  Arms: Natural Claim
Behavioral: Sugar Claim — Participants assigned to this condition will view three alcoholic beverages that carry the following claim: Zero sugar
  Arms: Sugar Claim
Behavioral: Fruit Claim — Participants assigned to this condition will view three alcoholic beverages that carry the following claim: Made with real fruit
  Arms: Fruit Claim

SUMMARY:
This study aims to examine the effects of marketing claims on alcoholic beverage packaging on alcohol consumers' perceptions and intentions. Participants will be randomized to view three images of alcoholic beverages (beer, hard seltzer, flavored malt beverage) with one of three marketing claims (or a no claim control), and then queried about their perceptions of the product and intentions to consume the product.

DETAILED DESCRIPTION:
This study aims to assess whether exposure to common marketing claims on alcoholic beverages impact alcohol consumer's perceptions of and intentions to consume the product. We aim to enroll approximately 1,500 adults ages 21 years and older who have consumed alcohol in the past year.

This study will be conducted online. After providing informed consent, participants will be randomly assigned to one of four conditions: either one of three marketing claims, or a no-claim control.

Participants view three alcohol products (beer, hard seltzer, and flavored malt beverage) in a random order within their assigned condition. After viewing each product, they will respond to survey items assessing their perceptions and intentions to consume the product.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 21 years and older
* Consumed alcohol at least once in the last year
* Able to complete a survey in English

Exclusion Criteria:

- Not living in the US

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-09-17 (Estimated); Study Completion 2026-09-17 (Estimated)

PRIMARY OUTCOMES:
Openness to consume | Baseline
  Measured using four survey items: 1.) "How open are you to trying this drink in the next two weeks?" 2.) "How open are you to buying this drink in the next two weeks? " 3.) "How open are you to consuming one serving of this drink in the next two weeks? One serving of this product is one 12 ounce can or bottle." and 4.) "How open are you to drinking x servings of this drink in one sitting in the next two weeks?" where x = 4 if the participant's gender is female, 5 otherwise Response options are on a 5-point scale with lowest endorsement (Not at all open) coded as 1 and highest endorsement (Extremely open) coded as 5.

SECONDARY OUTCOMES:
Perceived healthfulness | Baseline
  Measured using the following survey item: "How healthy or unhealthy would it be for you to consume one serving of this drink per day?" Response options are on a 5-point scale ranging from "Very unhealthy", coded as 1 to "Very healthy", coded as 5.
Perceived alcohol content | Baseline
  Measured using the following survey item: "What percentage alcohol by volume (ABV) do you think this drink contains?" Response option will use a slider scale with values ranging from 0% to 100%.
Perceived calorie content | Baseline
  Measured using the following survey item: "How many calories do you think one serving of this drink contains?" Response option will be a free numeric response ranging from 0-700.
Cancer risk perceptions | Baseline
  Measured using the following survey item: "Indicate how much you disagree or agree with the following statement: Drinking this product would increase my risk of cancer." Response options are on a 5-point scale ranging from "Strongly disagree", coded as 1 to "Strongly agree", coded as 5.

CONTACTS AND LOCATIONS:
Overall Officials: Phoebe R Ruggles, MS, Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials